CLINICAL TRIAL: NCT04652414
Title: Corticosteroid Treatment for Community-Acquired Pneumonia to Improve Long-term Cognition: A Pilot Randomized Controlled Trial
Brief Title: Corticosteroids in Community Acquired Pneumonia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited enrollment due to the COVID-19 pandemic. Sponsor withdrew funding.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jin H. Han, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 200278
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Community-acquired Pneumonia; Cognition Disorder
MeSH Terms: conditions — Community-Acquired Pneumonia; Cognition Disorders | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Prednisone (Experimental): Patients randomized to the intervention arm will receive prednisone 50mg PO daily for 7 days.
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator): Patients will receive matching placebo PO daily for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Prednisone 50mg will be administered enterally for 7 days.
  Arms: Prednisone
Drug: Placebo — This is a matching placebo to prednisone.
  Arms: Placebo

SUMMARY:
This is a single-center, blinded, placebo-controlled pilot RCT evaluating corticosteroids for the treatment of Community Acquired Pneumonia (CAP) that will enroll 100 adults hospitalized with community-acquired pneumonia. The primary goal is to assess the feasibility of proposed trial procedures for use in a subsequent phase III trial powered on 6-month cognitive outcome (MOCA-Blind score). Key outcomes are six-month cognitive and functional status, duration and severity of symptoms, and mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years
2. Hospital admission to ward or ICU (including observation status admissions)
3. Acute pneumonia defined as fulfilling each of the following two criteria: (a) New (<7-day duration) or worsening symptoms consistent with a lower respiratory tract infection, including ≥ 1 of the following: cough, shortness of breath, chest pain, sputum production, or decline in mental status; (b) Radiographic findings on chest x-ray or CT consistent with acute pulmonary infection, including pulmonary opacities, infiltrates, or pleural effusion.
4. CRP ≥ 15 mg/dL within 24 hours of enrollment

Exclusion Criteria:

1. Systemic steroid use within the past 30-days.
2. Clinical team planning to treat with systemic steroids during this hospitalization independent of the study protocol.
3. Unable to randomize patient within 24 hours of hospital presentation.
4. Hospital-acquired pneumonia, defined as development of clinical and radiographic signs of pneumonia as an inpatient in an acute care hospital. (Residence in a nursing home or assisted living facility is not an exclusion criterion.)
5. Unable to follow simple commands or non-verbal prior to this acute illness.
6. Pre-existing severe dementia, defined as an Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) score ≥ 4.12.
7. Concomitant acute decompensated heart failure requiring intravenous diuretics
8. Serum sodium > 145 mEq/L (hypernatremia) or potassium < 3.5 mEq/L (hypokalemia) at screening and randomization
9. Systolic blood pressure > 180 mmHg or a diastolic blood pressure > 100 mmHg at the start and end of screening.
10. Any history of diabetes mellitus, having a serum blood glucose > 250 mg/dL, or requiring an anti-diabetic medication (e.g., insulin)
11. Previous allergic or adverse reaction to a corticosteroid
12. Severe immunosuppression, defined as any of the following: HIV with CD4 count < 200 cells/mm3, absolute neutrophil count < 500 cells/mm3, solid organ or hematopoietic stem cell transplant with in the past 90 days.
13. Cystic fibrosis
14. Active cancer, defined as new diagnosis or treatment for cancer in the past 6 months.
15. Any history of adrenal insufficiency
16. Substance abuse (alcohol, opioid, benzodiazepines, methamphetamines, cocaine) within the past year
17. Any history of hospitalizations due to psychiatric illnesses within the past year
18. Gastro-intestinal bleeding treated with hospital admission and/or blood transfusion within the past 3 months.
19. Pre-existing medical condition resulting in a life expectancy < 6 months.
20. Clinical team does not believe the patient should enter the study due to concerns about potential steroid-related complications.
21. Alternative non-pneumonia illness accounts for the acute clinical or radiographic findings that meet the study's inclusion criteria.
22. Unable to take the enteral study medicine by mouth or tube
23. Prior enrollment in this study at any time
24. Non-English speaking
25. Confirmed or suspected COVID-19 as the cause of the patient's acute illness -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Feasibility as determined by the number of subjects who are successfully recruited and complete follow-up | 1.5 years
  Feasibility will be defined as: (a) recruitment and successful protocol completion of 100 patients; (b) corticosteroids being well tolerated, as shown by similar severity and frequency of adverse events in the intervention and placebo groups; (c) successful completion of 6-month cognitive assessments by >80% of survivors; and (d) the primary cognitive outcome Montreal Cognitive Assessment-Blind (MOCA-Blind) numerically favoring the intervention group with the one-tailed upper 80% confidence interval of the difference in MOCA-Blind between the intervention and placebo groups containing the minimally-important clinical difference (2 points on the MOCA-Blind).

SECONDARY OUTCOMES:
Global cognition as measured by the Montreal Cognitive Assessment-Blind (MOCA-Blind) | 6-months
  This is a measure of global cognition based on the assessment of attention concentration, memory, language, conceptual thinking, calculations, and orientation. Scores range from 0 to 22 with higher scores indicating better cognition.
Severity of pneumonia symptoms as measured by the Community-Acquired Pneumonia Symptom (CAP-Sym) Questionnaire | 3-days
  This is a 18-item scale to determine the presence and severity of pneumonia symptoms. Each item is graded on a 6-point Likert scale. Scores range from 0 to 90 with higher scores indicating more severe symptoms.
Severity of pneumonia symptoms as measured by the Community-Acquired Pneumonia Symptom (CAP-Sym) Questionnaire | 7-days
  This is a 18-item scale to determine the presence and severity of pneumonia symptoms. Each item is graded on a 6-point Likert scale. Scores range from 0 to 90 with higher scores indicating more severe symptoms.
Severity of pneumonia symptoms as measured by the Community-Acquired Pneumonia Symptom (CAP-Sym) Questionnaire | 30-days
  This is a 18-item scale to determine the presence and severity of pneumonia symptoms. Each item is graded on a 6-point Likert scale. Scores range from 0 to 90 with higher scores indicating more severe symptoms.
Quality of life as measured by the EQ-5D-5L | 6-months
  Characterizes quality of life and contains 5-dimensions ("5D") related to everyday living: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. It asks patients to rate their current global health status from 0 (worst health you can imagine) to 100 (best health you can imagine). Scores range from -0.573 to 1.000 with higher scores indicating better quality of life.
Basic activities of daily living (ADL) as measured by the Barthel's Index | 6-months
  Quantifies pre-illness basic ADLs such as bathing, dressing, toileting, transferring, continence, and feeding. Scores range from 0 to 20 with higher scores indicating better functioning.
Instrumental ADL as measured by Lawton Instrumental Activities of Daily Living Scale (IADLs) | 6-months
  Quantifies pre-illness IADLs - ability to use the phone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and finances. Scores range from 0 to 8 with higher scores indicating better functioning.
Employment status as characterized by the Outcomes After Critical Illness and Surgery (OACIS) Employment Status Questionnaire | 6-months
  9-item survey that characterizes the patient's baseline (prior to the critical illness) and current level of employment (full, partial, or not employed). Patients will be categorized as loss of employment or no loss of employment.
Vital status (dead / alive) | Baseline to hospital discharge, approximately 5 days
  Death during the index hospitalization will be recorded.
Vital status (dead / alive) | 6-months
  Death within 6-months will be recorded.
Intensive care unit admission (yes/no) | Baseline to hospital discharge, approximately 5 days
  Intensive care unit admission at any point during the index hospitalization will be recorded.
Mechanical ventilation (yes/no) | Baseline to hospital discharge, approximately 5 days
  Invasive mechanical ventilation is defined as new assisted positive pressure breathing through an endotracheal tube or tracheostomy for any duration. Noninvasive ventilation through a mask or nasal prongs does not satisfy the outcome of invasive mechanical ventilation.
Vasopressor use (yes/no) | Baseline to hospital discharge, approximately 5 days
  defined as the administration of any of the following medications by continuous infusion for at least 1 hour during the index hospitalization: norepinephrine, epinephrine, dopamine, phenylephrine or vasopressin.
Pleural drainage (yes/no) | Baseline to hospital discharge, approximately 5 days
  Pleural drainage is defined as removal of fluid from the pleural space by any procedure at the bedside or in the operating room during the index hospitalization; procedures such as thoracentesis and video-assisted thorascopic surgery (VATS) may be used to drain pleural fluid.
Hospital length of stay in (days) | Baseline to hospital discharge, approximately 5 days
  Duration of hospitalization (presentation to hospital discharge) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Han, MD,MSc, Principal Investigator — Vanderbilt University Medical Center; Wesley Self, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No